CLINICAL TRIAL: NCT00071253
Title: A Randomized, Double-Blind Study of Depakote Monotherapy, Olanzapine Monotherapy, and Combination Therapy of Depakote Plus Olanzapine in Stable Subjects During the Maintenance Phase of Bipolar Illness
Brief Title: Depakote Monotherapy, Olanzapine Monotherapy, and Combination Therapy of Depakote Plus Olanzapine in Stable Subjects During the Maintenance Phase of Bipolar Illness
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Abbott (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M02-551
Record Dates: First submitted 2003-10-16; First posted 2003-10-20 (Estimated); Last update posted 2006-08-04 (Estimated); Status verified 2006-08

CONDITIONS: Bipolar Disorder
Keywords: Bipolar Disorder - Mania
MeSH Terms: conditions — Bipolar Disorder | interventions — Valproic Acid; Olanzapine

INTERVENTIONS:
Drug: Divalproex Sodium (Delayed-Release Tablets)
Drug: Divalproex Sodium (Extended-Release Tablets)
Drug: Olanzapine

SUMMARY:
The purpose of this study is to assess the efficacy and safety of continued combination therapy using Depakote plus olanzapine, vs. Depakote monotherapy and olanzapine monotherapy in stable subjects during the maintenance phase of bipolar illness.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV-TR primary diagnosis of Bipolar I Disorder as confirmed by the SCID
* Outpatient receiving treatment with a combination of Depakote plus olanzapine for their bipolar illness and considered clinically stable (e.g., no more than minimal symptoms, no psychiatric hospitalizations, no increase in intensity of clinical interventions) for the preceding 4 months
* Identified at Screening a most bothersome side effect listed in the UKU which makes switching to monotherapy desirable
* MRS total score < 12 on two consecutive ratings, separated by at least 5 days (Screening and Day 1)
* DSS score < 13 on two consecutive ratings, separated by at least five days (Screening and Day 1)
* CGI-S score < 3 on two consecutive ratings, separated by at least five days (Screening and Day 1)
* Serum valproate level > 45 mcg/mL, and a maximum allowable dose of Depakote of 3000 mg/day at Screening
* Olanzapine dose between 5 and 20 mg/day at Screening

Exclusion Criteria:

* History of schizophrenia or schizoaffective disorder
* Axis I (e.g., anxiety disorder) or Axis II (e.g., personality disorder) that would interfere with compliance or confound interpretation of study results
* Has taken antipsychotics, mood stabilizers, or anticonvulsants (unless specifically for seizure control) other than Depakote or olanzapine in the four months prior to randomization. Other psychotropics (e.g., antidepressants, anxiolytics) with the exception of stimulants, that have been used routinely to maintain stability in the preceding four months may be continued, but not increased or decreased
* Has first manic episode after age 60
* Has ever taken clozapine
* Has received depot neuroleptic medication within six months of randomization
* Urine toxicology screen is positive for phencyclidine (PCP), opiates, cocaine or amphetamines
* History of active alcohol or substance abuse/dependence within 90 days prior to Screening
* Known history of non-response to either Depakote or olanzapine monotherapy for the treatment of bipolar disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180
Dates: Start 2003-07

PRIMARY OUTCOMES:
CGI-s
CGI-i
MRS
DSS
SADS-C

CONTACTS AND LOCATIONS:
Overall Officials: Global Medical Information, Study Director — Abbott
Locations (15):
- United States (15):
  - Behavioral and Medical Research, LLC, Anaheim, California
  - Synergy Clinical Research, Chula Vista, California
  - Clinical Trial Management, Fort Meyers, Florida
  - Segal Institute for Clinical Research, North Miami, Florida
  - Rush Presbyterian - St. Luke's, Chicago, Illinois
  - University of Louisville Outpatient Psychiatry, Louisville, Kentucky
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Creighton University Department of Psychiatry, Omaha, Nebraska
  - Lake Mead Hospital, North Las Vegas, Nevada
  - NYU School of Medicine, New York, New York
  - University Hospital of Cleveland, Cleveland, Ohio
  - R. Ranjan, MD & Associates, Inc., Lyndhurst, Ohio
  - IPS Research, Oklahoma City, Oklahoma
  - UTMB Dept. of Psychiatry, Galveston, Texas
  - Zablocki VAMC, Milwaukee, Wisconsin